CLINICAL TRIAL: NCT04130178
Title: Nerve Block of the Proximal Interphalyngeal Joints PIPs in Rheumatoid Arthritis (RA) Patients: a Prospective Pilot Study
Brief Title: Nerve Block of the Proximal Interphalangeal Joints PIPs in Rheumatoid Arthritis (RA) Patients: a Prospective Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahrous, Associate professor, Sohag University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 4/10/2019
Record Dates: First submitted 2019-10-11; First posted 2019-10-17 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Nerve Block; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacine injected (Active Comparator): Half ml of Bupivicaine hydrochloride .5% (Marcaine, Pfizer) was injected through a 27G needle at the level of the volar proximal digital crease of the 2nd and 3rd PIP on each side of the selected joint.
  Interventions: Drug: Nerve block
- Control group (Placebo Comparator): Saline was injected subcutaneously in the 2nd and 3rd PIP on each side of the selected joint.
  Interventions: Drug: Saline injection

INTERVENTIONS:
Drug: Nerve block — block of the digital nerves in rheumatoid arthritis patient
  Arms: Bupivacine injected
Drug: Saline injection — subcutaneous saline injection
  Arms: Control group

SUMMARY:
Researchers will include 83 rheumatoid arthritis patients (either early or established) diagnosed after 2010 ACR/EULAR criteria with bilateral hand arthritis aged 18 or above. Nerve block to the neural bundle of the 2nd and 3rd PIPs will be done to one hand (the dominant in half of the participants and the non-dominant in the remaining). The other hand will be used as a control and injected subcutaneously with saline. Half ml of Bupivacaine will be injected through a 27G needle at the level of the volar proximal digital crease of the 2nd and 3rd PIP. The needle will be directed alternatively toward the two pedicles on both sides.

PIPs of the 2nd and 3rd fingers in both hands will be examined EULAR-OMERACT scoring system at 0, 2 weeks, and 2 months intervals. Visual analog scale (VAS) for each hand will be used at the same intervals. There are no certain conditions for medications and all the patients were using sDMARDS.

DETAILED DESCRIPTION:
PIPs of the 2nd and 3rd fingers at the control group will be injected with .5 mL of saline on each joint through a 27G needle.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis patient according to ACR/EULAR criteria
* age >18
* bilateral hand affection

Exclusion Criteria:

* peripheral neuropathy
* other chronic arthritis
* patient who did mastectomy or any other hand operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
Change in pain | 0 time after 2 weeks and after 2 months
  by visual analogue sclae
Change in the degree of inflammation | at 0 time after 2 weeks and after 2 months
  Musculoskeletal ultrasound evaluation by EULAR-OMERACT score

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elsaman, PhD, Principal Investigator — Sohag University
Locations (1):
- Sohag university, Sohag, Egypt